CLINICAL TRIAL: NCT05421039
Title: Unintended Home Injuries in Under-5 Children in Sohag Governorate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Gamal Salem, Unintended Home Injuries in Under-5 Children in Sohag Governorate, Sohag University
Other Study IDs: Soh-med-22-06-02
Record Dates: First submitted 2022-06-12; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Unintended Home Injuries in Under-5 Children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Group (1): With the exposure
  Interventions: Behavioral: Exposure to unintended injuries
- Group (2): Without the exposure

INTERVENTIONS:
Behavioral: Exposure to unintended injuries — After taking a verbal consent , an explanation of the study will be given to the caregivers
  , those who fulfill the inclusion criteria will be enrolled in the study. Personal interviews by the researcher will be made with individuals or groups (2-4 persons) , participants will be chosen by means of systematic random sampling among visitors ؛ every 3rd or 5th child according to density and flow of attendance .
  the investigator will fill the questionnaire through personal interview with the caregivers
  Groups: Group (1)

SUMMARY:
Child injuries are a major public health problem . Globally, unintended injury is one of the top 15 causes of death across all age groups of children aged؛ 0-19 years, In children under the age of five, the majority of injuries occur in the home.

Injuries is a health concern in every country around the world, affecting both developed and developing countries, causing over 5.8 million deaths per year or 15,000 deaths per day .

A WHO surveillance study conducted in four developing countries showed that Egypt had a prevalence of 32 % of childhood injuries which was the highest one .

The home is the place where children spend most of their time, the home environment is the most common place for childhood injuries

DETAILED DESCRIPTION:
There is a lack of studies related to unintended home injuries in under-5 children in Sohag Governorate , unintended home injuries may result in temporary or permanent disability and requires medical attention and continuous care .

A limited number of child home injuries lead to hospitalization , so hospital based studies may ignore small scale injuries which couldn't be registered.

Unintended home injuries may influence health, education, and family economy of the affected children.

Unintended home injuries is one of the preventable causes of child morbidity and mortality , so we should know the prevalence and factors predisposing to it .

The aim of the study is to decrease morbidities and mortalities associated with unintended home injuries in under-5 children in Sohag Governorate by assessing prevalence and epidemiology of unintended home injuries in under-5 children in Sohag Governorate ,measuring extent of morbidities and mortalities associated with unintended home injuries in under-5 children in Sohag Governorate , determining factors predisposing to unintended home injuries in under-5 children in Sohag Governorate .

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted through personal interview with caregivers of under-5 children who accept to participate in it .

Exclusion Criteria:

* Caregivers who refuse to participate in the study and caregivers of children who experienced intended home injuries will be excluded from the study.

Ages: 2 Months to 5 Years | Sex: All
Age Groups: Child
Study Population: The study targeted under-5 children with their caregivers
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Unintended Home Injuries in Under-5 Children in Sohag Governorate | 2 months
  Assess prevalence and epidemiology of unintended home injuries in under-5 children in Sohag Governorate
Unintended Home Injuries in Under-5 Children in Sohag Governorate | 2 months
  Measure extent of morbidities and mortalities associated with unintended home injuries in under-5 children in Sohag Governorate .
Unintended Home Injuries in Under-5 Children in Sohag Governorate | 2 months
  Determine factors predisposing to unintended home injuries in under-5 children in Sohag Governorate .

IPD SHARING:
Plan to Share IPD: Undecided